CLINICAL TRIAL: NCT06191276
Title: Combating Hospital-related Function Decline Among Prefrail Older Adults: Pilot Testing of a Strength-based Tailored-Exercise Program at Home (STEP@Home)
Brief Title: Combating Hospital-related Function Decline Among Prefrail Older Adults: A Pilot Study
Acronym: STEP@Home
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Yu, Doris Sau Fung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STEP@Home
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Frailty; Geriatrics
Keywords: Geriatric patients; hospitalization-associated functional decline (HAFD); Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STEP@Home Intervention (Experimental): This arm involves participants undergoing the 20-week STEP@Home multi-component exercise training program. The program is designed to recondition the functional status of older adults in the post-discharge period and develop long-term exercise engagement.
  Interventions: Behavioral: STEP@Home Intervention
- Usual care (Active Comparator): Participants in this group receive the usual post-discharge care provided in the hospital setting, including general education on medication, disease-related self-care, and regular medical follow-ups.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: STEP@Home Intervention — STEP@Home is a multi-component exercise program designed for prefrail older adults that incorporates active strategies to promote long-term engagement. The optimal level of training is 45-60 minutes of exercise three times per week for at least 20 weeks. For prefrailty management, emphasis is placed on balancing and resistance training (around 15-20 min each) to improve muscle strength and gross mobility and prevent falls. Aerobic and flexibility exercises (10 min each) are also included to improve fitness and walking pace. Sixteen training tasks, including but not limited to those recommended by Vivifrail, for each exercise component (namely, resistance, balance, flexibility and aerobic training) will be adopted. A training manual with step-by-step illustrations of each task in pictures and text will be provided to the subjects, together with a set of simple, easy-to-access equipment (water bottle, elastic band and weight-bearing belt) to support task fulfilment.
  Arms: STEP@Home Intervention
Behavioral: Usual care — Usual Care Activities will be provided by the elderly community center such as dementia or caregiver supporting service. They will be allowed to use the regular service provided such services are not related to physical activity or exercise training.
  Arms: Usual care

SUMMARY:
This study focuses on the "Strength-based Tailored-Exercise Program at Home (STEP@Home)" aimed at improving health outcomes for geriatric patients at risk of hospitalization-associated functional decline. It is a sequential mixed-method study that combines quantitative and qualitative approaches.

DETAILED DESCRIPTION:
The research is a pilot study to develop the STEP@Home intervention, integrating a strength-based, tailored exercise regimen for elderly patients post-hospital discharge. It addresses hospitalization-associated functional decline (HAFD) by engaging patients in sustainable self-practice of physical exercises at home. The study employs empowerment strategies, lifestyle-integrated functional exercises, and optimized tele-platform use to maximize therapeutic benefits. By focusing on empowering patients through sustainable self-practice of physical exercises at home, it aims to enhance physical functions and improve health-related quality of life. The study also has significant real-world implications, potentially offering a scalable, effective solution for the broader geriatric population to manage HAFD, thereby reducing healthcare costs and improving overall well-being. The research intends to assess the program's impact on physical functions and health-related quality of life, utilizing a sequential mixed-method approach for a comprehensive evaluation.

ELIGIBILITY:
Inclusion Criteria:

* i) aged 60 or above, ii) prefrail as defined by a score of 1-2 on the Frail Scale (FS) which measures fatigue, resistance, ambulation, illness and weight loss over the last 4 weeks, iii) discharged home without any community care referral, iv) cognitively capable to receive exercise training as indicated by an Abbreviated Mental Test score of ≥ 6, and v) consented to participate

Exclusion Criteria:

* (i) engaging in moderate or vigorous exercise (>60min/week) in the past 6 months, and (ii) with conditions contradictory to exercise training (e.g., acute muscular-skeletal problem, acute and unstable cardio-respiratory disease, etc).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The 5-item FRAIL Scale (FS) | Baseline
  measuring frailty status based on the five phenotypes including fatigue, resistance, ambulation, illness and recent weight loss. With one point assigned to each phenotype, a total score of 0 indicates 'robust,' 1-2 'prefrail' and 3-5 'frail' with good validity.
The 5-item FRAIL Scale (FS) | 10th week
  measuring frailty status based on the five phenotypes including fatigue, resistance, ambulation, illness and recent weight loss. With one point assigned to each phenotype, a total score of 0 indicates 'robust,' 1-2 'prefrail' and 3-5 'frail' with good validity.
The 5-item FRAIL Scale (FS) | 20th week
  measuring frailty status based on the five phenotypes including fatigue, resistance, ambulation, illness and recent weight loss. With one point assigned to each phenotype, a total score of 0 indicates 'robust,' 1-2 'prefrail' and 3-5 'frail' with good validity.
The 5-item FRAIL Scale (FS) | 28th week
  measuring frailty status based on the five phenotypes including fatigue, resistance, ambulation, illness and recent weight loss. With one point assigned to each phenotype, a total score of 0 indicates 'robust,' 1-2 'prefrail' and 3-5 'frail' with good validity.
The 11-item Edmonton Frail Scale | Baseline
  supplementing the FS by providing more comprehensive coverage to capture frailty severity (e.g., functional independence and performance, general health status, mood) on a continuous scale.
The 11-item Edmonton Frail Scale | 10th week
  supplementing the FS by providing more comprehensive coverage to capture frailty severity (e.g., functional independence and performance, general health status, mood) on a continuous scale.
The 11-item Edmonton Frail Scale | 20th week
  supplementing the FS by providing more comprehensive coverage to capture frailty severity (e.g., functional independence and performance, general health status, mood) on a continuous scale.
The 11-item Edmonton Frail Scale | 28th week
  supplementing the FS by providing more comprehensive coverage to capture frailty severity (e.g., functional independence and performance, general health status, mood) on a continuous scale.
The Short Physical Performance Battery (SPPB) | Baseline
  combing a balance test, gait velocity and chair stand to reflect the functional capacity of older adults.21 Its score range is 0-12 in an ascending trend toward increased functional status.The SPPB has good predictive validity against functional decline, rehospitalization and mortality in older adults.
The Short Physical Performance Battery (SPPB) | 10th week
  combing a balance test, gait velocity and chair stand to reflect the functional capacity of older adults.21 Its score range is 0-12 in an ascending trend toward increased functional status.The SPPB has good predictive validity against functional decline, rehospitalization and mortality in older adults.
The Short Physical Performance Battery (SPPB) | 20th week
  combing a balance test, gait velocity and chair stand to reflect the functional capacity of older adults.21 Its score range is 0-12 in an ascending trend toward increased functional status.The SPPB has good predictive validity against functional decline, rehospitalization and mortality in older adults.
The Short Physical Performance Battery (SPPB) | 28th week
  combing a balance test, gait velocity and chair stand to reflect the functional capacity of older adults.21 Its score range is 0-12 in an ascending trend toward increased functional status.The SPPB has good predictive validity against functional decline, rehospitalization and mortality in older adults.

SECONDARY OUTCOMES:
The Life Space Assessment (LSA-C) | Baseline
  capturing mobility level of relatively independent prefrail older adults in everyday activities. It assesses the level of mobility at five life-space levels in the past 4 weeks: living room other than the bedroom, ii) outside the house, iii) the neighborhood (within 800m of home), iv) outside the neighborhood (within 8km) and v) outside the town (beyond 16km). Example locations representing various distances from subjects' homes will be provided to facilitate the responses. The LSA-C has reliability of 0.88, with good criterion and construct validity.
The Life Space Assessment (LSA-C) | 10th week
  capturing mobility level of relatively independent prefrail older adults in everyday activities. It assesses the level of mobility at five life-space levels in the past 4 weeks: living room other than the bedroom, ii) outside the house, iii) the neighborhood (within 800m of home), iv) outside the neighborhood (within 8km) and v) outside the town (beyond 16km). Example locations representing various distances from subjects' homes will be provided to facilitate the responses. The LSA-C has reliability of 0.88, with good criterion and construct validity.
The Life Space Assessment (LSA-C) | 20th week
  capturing mobility level of relatively independent prefrail older adults in everyday activities. It assesses the level of mobility at five life-space levels in the past 4 weeks: living room other than the bedroom, ii) outside the house, iii) the neighborhood (within 800m of home), iv) outside the neighborhood (within 8km) and v) outside the town (beyond 16km). Example locations representing various distances from subjects' homes will be provided to facilitate the responses. The LSA-C has reliability of 0.88, with good criterion and construct validity.
The Life Space Assessment (LSA-C) | 28th week
  capturing mobility level of relatively independent prefrail older adults in everyday activities. It assesses the level of mobility at five life-space levels in the past 4 weeks: living room other than the bedroom, ii) outside the house, iii) the neighborhood (within 800m of home), iv) outside the neighborhood (within 8km) and v) outside the town (beyond 16km). Example locations representing various distances from subjects' homes will be provided to facilitate the responses. The LSA-C has reliability of 0.88, with good criterion and construct validity.
European Quality of Life 5 Dimensions 5 Level Version (EuroQoL-5D-5L) | Baseline
  assessing Health-Related Quality of Life and generating the utility score for Cost-Effectiveness Analysis. It comprises a 5-level response set (5-L), including mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a 0-100 visual analogue scale to measure perceived health.
European Quality of Life 5 Dimensions 5 Level Version (EuroQoL-5D-5L) | 10th week
  assessing Health-Related Quality of Life and generating the utility score for Cost-Effectiveness Analysis. It comprises a 5-level response set (5-L), including mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a 0-100 visual analogue scale to measure perceived health.
European Quality of Life 5 Dimensions 5 Level Version (EuroQoL-5D-5L) | 20th week
  assessing Health-Related Quality of Life and generating the utility score for Cost-Effectiveness Analysis. It comprises a 5-level response set (5-L), including mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a 0-100 visual analogue scale to measure perceived health.
European Quality of Life 5 Dimensions 5 Level Version (EuroQoL-5D-5L) | 28th week
  assessing Health-Related Quality of Life and generating the utility score for Cost-Effectiveness Analysis. It comprises a 5-level response set (5-L), including mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a 0-100 visual analogue scale to measure perceived health.
Unplanned hospital readmissions | Baseline
  will be monitored for a period of 32 weeks via the Hospital Authority Clinical Management System. Information on the date of admission, total length of stay and index diagnosis of admission will be retrieved. The research nurse will also ask the subjects about admissions to private hospitals.
Unplanned hospital readmissions | 10th week
  will be monitored for a period of 32 weeks via the Hospital Authority Clinical Management System. Information on the date of admission, total length of stay and index diagnosis of admission will be retrieved. The research nurse will also ask the subjects about admissions to private hospitals.
Unplanned hospital readmissions | 20th week
  will be monitored for a period of 32 weeks via the Hospital Authority Clinical Management System. Information on the date of admission, total length of stay and index diagnosis of admission will be retrieved. The research nurse will also ask the subjects about admissions to private hospitals.
Unplanned hospital readmissions | 28th week
  will be monitored for a period of 32 weeks via the Hospital Authority Clinical Management System. Information on the date of admission, total length of stay and index diagnosis of admission will be retrieved. The research nurse will also ask the subjects about admissions to private hospitals.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Sau Fung YU, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Alice Ho Miu Ling Nethersole Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Only study investigators and research assistants involved in the study will have access to the data.